CLINICAL TRIAL: NCT06177015
Title: Randomized Controlled Study on the Efficacy and Safety of Intermittent Darolutamide Treatment in the Triple Therapy of Metastatic Hormone Sensitive Prostate Cancer
Brief Title: Intermittent Darolutamide Treatment in the Triple Therapy of mHSPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hua Lixin, M.D., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-662
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Prostate Cancer; Intermitent Anti-androgen Therapy
Keywords: triple treatment regimen; mHPSC; Darolutemide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Intervention Model Description: Two independent arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous treatment group (Active Comparator): Darolutamide: 600mg, bid+ADT: Leuprorelin (3.6mg qm or 10.8mg q3m) or goserelin 80mg qm until mCRPC
  Interventions: Drug: Darolutamide continuous
- Intermittent treatment group (Experimental): Only ADT as background treatment without Darolutamide. PSA check every three months, when the patient's PSA > 1ng/ml (or PSA > 1ng/ml and PSA has risen by more than 20% comparing baseline), restart the darolutamide, until mCRPC.
  Interventions: Drug: Darolutamide intermittent

INTERVENTIONS:
Drug: Darolutamide continuous — standard of care
  Other Names: Darolutamide
  Arms: Continuous treatment group
Drug: Darolutamide intermittent — experimental group
  Other Names: Darolutamide
  Arms: Intermittent treatment group

SUMMARY:
To evaluate the efficacy and safety of intermittent use of darolutamide compared to long-term use in combination with ADT and docetaxel in the treatment of mHSPC patients.

DETAILED DESCRIPTION:
Patients will firstly receive 6 months of darolutamide in combination with docetaxel and ADT treatment.

1. When the patient reaches:

1. PSA ≤ 0.2ng/ml
2. Or PSA > 0.2ng/ml but with more that 90% decrease comparing baseline
3. Without newly discovered metastatic lesions. They will be randomly assigned in a 1:1 ratio to either continuous treatment group or intermittent treatment group (1) Continuous treatment group: Darolutamide: 600mg, bid+ADT: Leuprorelin (3.6mg qm or 10.8mg q3m) or goserelin 80mg qm until mCRPC; (2) Intermittent treatment group: Only ADT as background treatment without Darolutamide. PSA check every three months, when the patient's PSA > 1ng/ml (or PSA > 1ng/ml and PSA has risen by more than 20% comparing baseline), restart the darolutamide, until mCRPC.

2. When the patient:

1. PSA > 0.2ng/ml and has not decreased by 90% compared to baseline
2. Or has new metastatic lesions, they will exit the study. Imaging assessment will be conducted every 3 months

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for this study:

1. Male aged ≥18 years;
2. Histologically or cytologically confirmed prostate adenocarcinoma;
3. Metastatic disease (confirmed by conventional imaging);
4. ECOG performance status of 0-1;
5. Suitable for ADT and docetaxel treatment;
6. Good bone marrow, kidney, and liver function:

1. (1) Hematological examination (no blood transfusion or use of hematopoietic growth factors within 7 days before screening):

1. Hemoglobin (HB) ≥ 90g/L; 2. Absolute neutrophil count (ANC) ≥ 1.5×109/L; 3. Platelets (PLT) ≥ 80×109/L; 2. (2) Blood biochemistry examination (no blood transfusion or albumin within 7 days before screening):

1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN
2. Total bilirubin (TBIL) ≤ 2.0 × ULN;
3. Serum creatinine (Cr) ≤ 2.0×ULN;

7. Willing to participate in this study, sign an informed consent form, and have good compliance

Exclusion Criteria:

1. No metastatic disease;
2. Prior treatment with: a) Second-generation ARis or other experimental ARis b) CYP17 enzyme inhibitors such as abiraterone acetate or oral ketoconazole for anti-tumor treatment of prostate cancer c) Chemotherapy or immunotherapy prior to randomization for prostate cancer
3. Received radiotherapy within 2 weeks before starting 6 months of darolutamide + docetaxel + ADT treatment;
4. Stroke, myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass surgery, congestive heart failure (New York Heart Association class III or IV);
5. History of malignant tumors;
6. Planned receipt of other anti-tumor treatment during the study treatment period;
7. Known allergy to the above drug components;
8. Difficulty swallowing, chronic diarrhea, intestinal obstruction, and various factors affecting drug intake and absorption;
9. Refusal to sign the informed consent form;
10. Investigator's opinion that the participant is not suitable for inclusion.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival | 36 months
  rPFS
Overall Survival | 36 months
  OS

SECONDARY OUTCOMES:
Time to castration-resistant prostate cancer | 36 months
  Time to mCRPC
Time to pain progression | through study completion, an average of 3 year
  TTPP

CONTACTS AND LOCATIONS:
Overall Officials: Lixxin Hua, Principal Investigator — Urology Dpt, First Affiliated Hospital of Nanjing Medical University
Locations (1):
- Urology dpt, First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT06177015/Prot_ICF_000.pdf